CLINICAL TRIAL: NCT06016361
Title: Evaluation of a Novel Amino Acid Based Moisturizing Cream as Part of the Daily Standard Skincare Regimen Recommended During Radiation Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Entrinsic Bioscience Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PR-23809
Record Dates: First submitted 2023-08-09; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Erythema; Radiation Therapy, Secondary Skin Reactions
MeSH Terms: conditions — Erythema | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Sham Comparator): Standard of Care
  Interventions: Other: Standard of care
- Investigational Product (Active Comparator): Investigational product
  Interventions: Other: VS-200Cr

INTERVENTIONS:
Other: VS-200Cr — Topical cream with moisturizing factors.
  Arms: Investigational Product
Other: Standard of care — AAD recommended course of care.
  Arms: Standard of Care

SUMMARY:
The goal of this clinical study is to evaluate a novel amino acid based moisturizing cream as part of the daily standard skincare regimen recommended during radiation therapy. The main aim of this study is to assess if the investigational product can improve skin redness associated with radiation therapy. Participants will apply a moisturizer daily during the course of their prescribed radiation therapy for breast cancer. Researchers will compare against the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Aged over 18 years old.
* Has been diagnosed with breast cancer and prescribed radiotherapy as a part of their cancer treatment.
* Planned radiotherapy, as prescribed by the oncologist, is expected to provide a total radiation dose of up to 60 gray within the first 4 weeks of treatment.
* Be able to adhere to proposed daily wound/site care as proposed by the protocol in line with the AADs recommendations.

Exclusion Criteria:

* Pre-existing skin conditions which in the opinion of the investigator could impact on the integrity of the study or compromise the safety of the patient (i.e., active eczema, psoriasis, or an open wound over the planned site of radiation).
* Have a concurrent medical condition or poor functional baseline which in the opinion of the investigator would make them unsuitable or able to fully comply with the study protocol.
* Are pregnant or actively breast feeding.
* Known allergic reactions to ingredients of the Investigational Product or the Standard of Care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-09-18 (Estimated); Primary Completion 2024-03-18 (Estimated); Study Completion 2024-03-18 (Estimated)

PRIMARY OUTCOMES:
Reduction in Erythema | Up to 12 weeks
  Evaluation of skin redness (both severity and size) with ScarletRed technology

CONTACTS AND LOCATIONS:
Locations (1):
- Advocate Radiation Oncology, Fort Myers, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided